CLINICAL TRIAL: NCT01917409
Title: Comparison of Conventional Laryngoscopy and Video-stylet to Assist Nasotracheal Intubation for Patients Undergoing Oro-Maxillo-facial Surgery
Brief Title: Video-stylet for Nasotracheal Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUH-IRB-20120320
Record Dates: First submitted 2013-07-10; First posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-07

CONDITIONS: Intubation, Difficult
Keywords: Conventional Laryngoscopy ,; Video-stylet ,; Nasotracheal Intubation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional laryngoscopy (Experimental): experimental conventional laryngoscopy group: laryngoscope is used to assist for nasotracheal intubation.
  Interventions: Device: conventional laryngoscopy
- video-stylet (Experimental): experimental video-stylet group:video-stylet is used to guide nasotracheal tube into trachea
  Interventions: Device: video-stylet

INTERVENTIONS:
Device: conventional laryngoscopy — the device is to assist nasotracheal intubation
  Other Names: Macintoish laryngoscope
  Arms: conventional laryngoscopy
Device: video-stylet — the device is to guide the nasotracheal tube into trachea
  Other Names: The Clarus Video System
  Arms: video-stylet

SUMMARY:
The purpose of this study is to compare conventional laryngoscopy with video-stylet (Trachway) for nasotracheal intubation in patients undergoing oro-maxillo-facial surgery.

ELIGIBILITY:
Inclusion Criteria:

1. patients with American Society of Anesthesiologists physical status I-III
2. aged 20-65 years
3. Requiring Nasotracheal Intubation under general anesthesia
4. unlimited mouth open
5. unlimited neck motion

Exclusion Criteria:

1. mouth open < 3 cm
2. Ankylosing arthritis patients.
3. BMI≧35 kg/m2

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
number of the patients with successful nasotracheal intubation and scoring difficult intubation scale | half an hour
  Nasotracheal intubation assisted by a video-stylet may be performed in patients undergoing oro-maxillo-facial surgery following induction of anesthesia (fentanyl 2 micro-gram/kg, thiamylal 5 mg/kg, cis-atracurium 0.2 mg/kg and propofol 1 mg/kg)

SECONDARY OUTCOMES:
time to intubate | 10 minutes
  time of Intubating the nasotracheal tube (NT) from selected nostril to trachea is continuously calculated but separately into two parts. part one: from termination of mask ventilation and mask removed from face, to the NT tip on the nasopharynx. part two: advancing NT from nasopharynx, through vocal cord into trachea, to present of 3 end tidal carbon dioxide waveforms.

OTHER OUTCOMES:
postoperative nasal bleeding, sore throat and hoarseness | 2 days
  Events of intubating related nasal bleeding are recorded on selected nostril and oral cavity at 3 minutes post-intubation and post-operatively. Incidences of sore throat and hoarseness are evaluated before patients out of recovery room and the following morning

CONTACTS AND LOCATIONS:
Overall Officials: Kuang I Cheng, MD., PhD., Study Director — Department of anesthesiology, Kaohsiung Medical University, Taiwan
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung, Taiwan

REFERENCES:
- [Derived] Hsu HT, Lin CH, Tseng KY, Shen YC, Chen CH, Chuang WM, Cheng KI. Trachway in assistance of nasotracheal intubation with a preformed nasotracheal tube in patients undergoing oral maxillofacial surgery. Br J Anaesth. 2014 Oct;113(4):720-1. doi: 10.1093/bja/aeu334. No abstract available. PMID 25236899